CLINICAL TRIAL: NCT06574997
Title: An Expanded Access Program for Retinitis Pigmentosa in Adults Aged 18 Years and Older
Brief Title: Expanded Access Program for RP in Adults
Status: Available | Type: Expanded Access
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Other Study IDs: OCU400-EAP
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; Modifier Gene Therapy; Modified Gene Therapy; RHO; RP; NR2E3; Subretinal Injection
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Drug: OCU400 — Participants will receive a subretinal injection of OCU400 modifier gene therapy product.

SUMMARY:
This intermediate-size patient population expanded access program is to provide access to investigational product OCU400 for up to 75 patients with Retinitis Pigmentosa (RP) outside of the ongoing clinical trial Phase 3 program for patients who do not have access to alternative Food and Drug Administration (FDA)-approved products for treatment of the disease.

DETAILED DESCRIPTION:
This expanded access protocol provides access to OCU400 for a subset of patients. Subjects will undergo specific ocular testing included in the study. Subjects will follow-up with physical examination, review of concomitant medication, blood work and ocular examinations for up to 52 weeks (about 12 months) post dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years of age at the time of informed consent.
2. Confirmed clinical and CLIA certified genetic diagnosis of RP (except subjects with AD-NR2E3 mutation)
3. Presence of photoreceptors as determined by spectral-domain optical coherence tomography (SD-OCT).

Exclusion Criteria:

1. Subject lacks evidence of outer nuclear layer, i.e., containing the nuclei of the retinal photoreceptors as determined by SD- OCT.
2. Considered unsuitable for any reason that may either place the subject at increased risk during participation or interfere with the interpretation of the study outcomes by the Investigator, or the Sponsor after reviewing the subject medical history and condition.
3. Previous treatment with a gene-therapy or cell therapy product, excluding OCU400.
4. Previous treatment with any investigational drug or device within one year, excluding OCU400.
5. Any contraindications for subretinal injection.
6. Cataract surgery within 3 months. YAG capsulotomy within 1 month. Any other intraocular surgery within 6 months

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Huma Qamar, MD, MPH, CMI, Study Chair — Ocugen
Locations (4):
- United States (4):
  - Associated Retina Consultants, Phoenix, Arizona
  - Advanced Research, Deerfield Beach, Florida
  - Erie Retina Research, Erie, Pennsylvania
  - Gundersen Health, La Crosse, Wisconsin